CLINICAL TRIAL: NCT00711217
Title: Evaluation of a Medical Food for Chronic Wounds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK15
Record Dates: First submitted 2008-06-23; First posted 2008-07-08 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-05

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- #1 Medical food (Experimental)
  Interventions: Other: Medical Food
- #2 Control (Placebo Comparator)
  Interventions: Other: Drink mix calorically similar to experimental product

INTERVENTIONS:
Other: Medical Food — twice daily
  Other Names: AN0806A
  Arms: #1 Medical food
Other: Drink mix calorically similar to experimental product — twice daily
  Other Names: AN0806B
  Arms: #2 Control

SUMMARY:
The study objective is to compare outcomes in subjects with a diabetic foot ulcer after 16 weeks of consuming a medical food versus a calorically similar control drink.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant
* diabetic
* neuropathic foot ulcer
* ABI> 0.7

Exclusion Criteria:

* uncontrolled DM
* collagen vascular disease or autoimmune disease
* wound infection; recent therapies with steroids
* growth factor or bioengineered tissue
* radiation therapy
* treatment with antibiotics within 1 week, Charcot's arthropathy of the foot
* active malignancy
* renal function impairment
* liver failure
* planned surgery
* myocardial infarction within 3 months
* malnutrition
* substance abuse
* taking conflicting oral nutritional supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Wound healing | 16 weeks

SECONDARY OUTCOMES:
QOL | 16 weeks
Wound healing measures | 16 weeks
Incidence of complications | 16 weeks
Clinical outcome data | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne Voss, PhD, RD, Study Director — Abbott Nutrition
Locations (51):
- United States (46):
  - University of Alabama, Birmingham, Alabama
  - Biomedical Research and Educational Foundation of Southern Arizona VA Health Care System, Tucson, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Foot and Ankle Specialist, Brawley, California
  - Center for Clinical Research, Inc, Castro Valley, California
  - Central Coast Foot and Ankle, Freedom, California
  - Foot and Ankle Clinic, Los Angeles, California
  - California School of Podiatric Medicine at Samuel Merritt University, Oakland, California
  - Therapeutics Clinical Research, San Diego, California
  - Advanced Clinical Research, San Jose, California
  - Pacific Wound Center, Stockton, California
  - Precision Foot and Ankle Centers - Torrance, Torrance, California
  - Diabetic Foot and Wound Center, Denver, Colorado
  - McHugh & Associates, Watertown, Connecticut
  - Doctor's Research Network, Miami, Florida
  - SCORE Physician Alliance, St. Petersburg, Florida
  - South Florida Wound Care Group, Tamarac, Florida
  - Ankle and Foot Associates, Temple Terrace, Florida
  - Aiyan Diabetes Center, Evans, Georgia
  - Garrett Noguchi, DPM, P.A., Honolulu, Hawaii
  - Rosalind Franklin University, Center for Lower Extremity Ambulatory Research, North Chicago, Illinois
  - Amputation Prevention Center Broadlawns Medical Center, Des Moines, Iowa
  - Christus Schumpert Wound Care Center & Hyperbaric Center, Shreveport, Louisiana
  - Chesapeake Research Group, Pasadena, Maryland
  - Foot Care, Endovascular and Vascular Services Boston University School of Medicine, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Harvard University, Boston, Massachusetts
  - American Center for Clinical Trials, Southfield, Michigan
  - Foot Healthcare Associates, Southfield, Michigan
  - Advance Foot & Ankle Center, Las Vegas, Nevada
  - VA Medical Center, Reno, Nevada
  - Gerard J. Furst, DPM, PLLC, Port Jefferson Station, New York
  - Akron General Medical Center, The Wound Care Center, Akron, Ohio
  - St. Vincent Charity Hospital, Wound Care Center, Cleveland, Ohio
  - ProMedica Health Systems, Toledo, Ohio
  - Blair Medical Associates, Inc., Altoona, Pennsylvania
  - Carlisle Regional Medical Center, Advanced Wound Healing Center, Carlisle, Pennsylvania
  - The Wound Institute and Research Center, Dunmore, Pennsylvania
  - Armstrong County Wound Healing Center, Kittanning, Pennsylvania
  - Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Limb Salvage Centre, Dallas, Texas
  - Complete Family Foot Care, McAllen, Texas
  - Robert Wunderlich, DPM, P.A., San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Trinity Mother Frances Hospitals and Clinics, Tyler, Texas
- Spain (2):
  - Clinica de Podologia, Ciudad Universitaria, Madrid
  - Centro de Diagnostico y Tratamiento Francisco Diaz, Madrid
- Chang Gung Memorial Hospital, Taipei, Taiwan
- United Kingdom (2):
  - Diabetic Foot Clinic, King's College Hospital, London
  - Manchester Diabetes Centre, Manchester